CLINICAL TRIAL: NCT02849756
Title: Future of the Older Patients After Intensive Care Unit
Acronym: DAAR
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0514
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Intensive Care Unit Syndrome
Keywords: Intensive care; elderly; autonomy; Future; older patients; intensive care unit
MeSH Terms: interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- older in intensive care unit: older (age superior at 85 years) hospitalized in intensive care unit. A follow-up until 6 months after hospitalization will determine the evolution of the quality of life and others secondary outcomes.
  Interventions: Other: older in intensive care unit

INTERVENTIONS:
Other: older in intensive care unit — It is an observational study with no intervention.

SUMMARY:
Estimate the future six months after the admission in an intensive care unit of the patients of 85 and more years old in terms of autonomy.

DETAILED DESCRIPTION:
The diverse studies published on the future of the elderly hospitalized in resuscitation place the limit very low, between 65 and 80 years. The feeling of a very bad forecast at these extreme ages pulls nevertheless a filter in the admission in ICU which has this day no scientific justification. The knowledge of the evolution after the hospitalization of these older patients can help to make certain decisions concerning as well the admission of these patients in ICU as the realization of invasive treatments.

After informal interrogation of numerous intensivists, it seems to take shape a bar around 85 years beyond which the forecast would be worse without more proof what consolidated the choice of this limit.

The reserved scores were already used in similar studies (simplified ALD).

Primary purpose :

* Describe the survival and the evolution of the quality of life after a stay in resuscitation for very old patients.
* The quality of life will be studied through a score of autonomy: the simplified ALD score.

The population will be described in general then by age bracket (more or less of 90 years old), according to the length of stay in ICU, the heavy treatments (artificial ventilation, renal replacement therapy) practiced, the initial gravity (score IGS 2). The impact of possible decisions of Limitation or Stop of Therapeutic Activates will also be taken into account.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 85 years old staying in intensive car units

Exclusion Criteria:

* Knaus D
* No possibly of call (phone) 6 months after ICU admission
* Patients who do not speak French
* Patients do not accept the participation

Min Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients older than 85 years hospitalized in intensive care unit will be included in this study.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
ALD score | Six month
  Geriatric score of autonomy

SECONDARY OUTCOMES:
survival | Six month
  survival

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Dr MICHEL, PH, Principal Investigator — René-Dubos Hospital
Locations (1):
- René-Dubos Hospital, Pontoise, Val d'Oise, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khouli H, Astua A, Dombrowski W, Ahmad F, Homel P, Shapiro J, Singh J, Nallamothu R, Mahbub H, Eden E, Delfiner J. Changes in health-related quality of life and factors predicting long-term outcomes in older adults admitted to intensive care units. Crit Care Med. 2011 Apr;39(4):731-7. doi: 10.1097/CCM.0b013e318208edf8. PMID 21263318
- [Background] Lewis-Newby M, Curtis JR, Martin DP, Engelberg RA. Measuring family satisfaction with care and quality of dying in the intensive care unit: does patient age matter? J Palliat Med. 2011 Dec;14(12):1284-90. doi: 10.1089/jpm.2011.0138. Epub 2011 Nov 22. PMID 22107108
- [Background] Biston P, Aldecoa C, Devriendt J, Madl C, Chochrad D, Vincent JL, De Backer D. Outcome of elderly patients with circulatory failure. Intensive Care Med. 2014 Jan;40(1):50-6. doi: 10.1007/s00134-013-3121-7. Epub 2013 Oct 17. PMID 24132383